CLINICAL TRIAL: NCT01819870
Title: A Randomized, Open-label, Multiple-dose, Crossover Phase I Study to Compare the Pharmacokinetic Characteristics and Safety of Dilatrend SR Capsule 32 mg and Dilatrend Tablet 25 mg in Healthy Male Subjects
Brief Title: Study to Compare the Pharmacokinetic Characteristics and Safety of Dilatrend SR Capsule 32mg and Dilatrend Tablet 25mg
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 125HPS12006
Record Dates: First submitted 2013-03-20; First posted 2013-03-28 (Estimated); Last update posted 2013-04-01 (Estimated); Status verified 2013-01

CONDITIONS: Essential Hypertension; Chronic Stable Angina; Congestive Heart Failure
Keywords: Carvedilol; Dilatrend SR capsule; Dilatrend Tablet; Pharmacokinetics; Healthy male subjects
MeSH Terms: conditions — Essential Hypertension; Angina, Stable; Heart Failure | interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dilatrend SR capsule 32mg (Experimental)
  Interventions: Drug: Dilatrend SR capsule 32mg
- Dilatrend IR tablet 25mg (Active Comparator)
  Interventions: Drug: Dilatrend IR tablet 25mg

INTERVENTIONS:
Drug: Dilatrend SR capsule 32mg — * 1 capsule, oral, once daily, 7days
  * over the period I&II(crossover)
  Arms: Dilatrend SR capsule 32mg
Drug: Dilatrend IR tablet 25mg — * 1 tablet, oral, once daily, 7days
  * over the period I&II(crossover)
  Arms: Dilatrend IR tablet 25mg

SUMMARY:
The purpose of this study is to compare the pharmacokinetic characteristics and safety of dilatrend SR capsule 32mg and Dilatrend tablet 25mg in healthy male subjects.

DETAILED DESCRIPTION:
Healthy male subjects are administrated multiple-dose over the period I and II (Crossover) of dilatrend SR capsule 32mg and dilatrend tablet 25mg.

ELIGIBILITY:
Inclusion Criteria:

* Between 20 aged and 35aged in healthy male
* Body Weight more than 50kg, and within 20% of ideal body weight(IBW).

  * IBW(kg) = {height(cm)-100}*0.9
* Have not any congenital or chronic disease and medical symptoms.
* Suitable results of inspections(laboratory test, ECG, etc) within 21 days before IP administration.
* Agreement with written informed consent

Exclusion Criteria:

* Subject has hypersensitivity reaction or clinically significant history about carvedilol or investigator drug.
* Clinically significant cardiovascular system, respiratory system, liver, kidney, endocrine system, gastrointestinal system, central nervous system, blood tumor, mental disease, skin disease, otorhinolaryngologic diseases and so on.
* Hypotension(SBP < 105mmHg or DBP < 65mmHg), Hypertension(SBP > 150mmHg or DBP > 100mmHg)
* Heart rate < 50times/minute
* Active liver disease or AST, ALT > 1.5*upper limit of normal range
* Creatinine clearance < 80mL/min
* Subject has a disease affecting drug's ADME or gastrointestinal surgery.
* Subject with symptoms of injured or acute disease within 28days before the first IP administration.
* Subject has a history of drug abuse or a positive reaction for drug abuse at the screening test for urine.
* Taking ETC medicine including oriental medicine within 14days before the first IP administration or Taking OTC medicine within 7days
* Subject takes an abnormal meal which affect the ADME of drug.
* Previously participate in other trial within 90days.
* Previously make whole blood donation within 60days or component blood donation within 30days before the first IP administration.
* Continued to be taking caffeine(caffeine > 5cup/day), drinking(alcohol > 21unit/week, 1unit = 10g = 12.5mL of pure alcohol) or during clinical trials can not be drunk or severe heavy smoker(cigarette > 10cigarettes/day).
* Subject with positive reaction about serum test(HBsAg, HCV Ab, HIV Ag/Ab, VDRL)
* Genetic problems such as galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption.
* An impossible one who participates in clinical trial by investigator's decision including for reason of laboratory test result.

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-05 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
In the steady state Dilatrend SR Capsule 32mg and Dilatrend tablet 25mg AUCtau | 0, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48hr post-dose (on last day of each period)
  AUCtau: Area under the plasma concentration-time curve for each dosing interval (from time 0 to 48 hours sample) determined using the linear trapezoidal rule

SECONDARY OUTCOMES:
In the steady state Dilatrend SR Capsule 32mg and Dilatrend tablet 25mg AUCinf | 0, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48hr post-dose (on last day of each period)
  AUCinf: Area Under the Concentration time curve with the last concentration extrapolated based on the elimination rate constant Kel
In the steady state Dilatrend SR Capsule 32mg and Dilatrend tablet 25mg Css,max | 0, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48hr post-dose (on last day of each period)
  Css,max : Maximum drug concentration in plasma determined directly from individual concentration-time data
In the steady state Dilatrend SR Capsule 32mg and Dilatrend tablet 25mg Css,min | 0, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48hr post-dose (on last day of each period)
  Css,min : Minimum drug concentration in plasma determined directly from individual concentration-time data
In the steady state Dilatrend SR Capsule 32mg and Dilatrend tablet 25mg Tss,max | 0, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48hr post-dose (on last day of each period)
  Tss,max : Time to reach maximum drug concentration in plasma calculated from [plasma] versus time profiles
In the steady state Dilatrend SR Capsule 32mg and Dilatrend tablet 25mg t½ | 0, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48hr post-dose (on last day of each period)
  t½ : Observed terminal elimination half-life
Number of participants with adverse events | From 1day to 37 days
  * Evaluated safety parameters included: physical examination, vital sign, laboratory test, ECG
  * adverse event monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Young-Ran Yoon, Principal Investigator — Kyungpook National University Hospital Clinical Trial Center
Locations (1):
- Kyungpook National University Hospital Clinical Trial Center, Daegu, Eok-dong 2(i)-ga Jung-gu, South Korea